



## Lung UltraSound as Alternative to Radiography after Thoracic Surgery (LUS-ART): a randomized controlled trial

Interim analysis summary

Date: 08-22-2024

Primary investigators: Sebastian Ullmark, Julia Jakobsson

Co-investigators: Emma Thorén, Joakim Engström

Sponsor: Laila Hellgren Johansson

Clinicaltrials.gov Identifier: NCT06261411

Swedish Ethical Review Authority Identifier: 2023-06510-01

Hospital/university trial Identifier: FOU2024-00038

## Contact information:

Dept. of Cardiothoracic surgery and -anaesthesia Uppsala University Hospital SE-751 85, Uppsala, SWEDEN sebastian.ullmark@uu.se



| Patient and perioperative characteristics | LUS (n=18) | CXR (n=24) | |
|---|---|---|---|
| Sex (no females, %) | 10 (55) | 16 (66) | 0.4631 |
| Age (yrs) | 66 (58 to 73) | 72 (67 to 76) | 0.1167 |
| BMI (kg m <sup>-2</sup> ) | 27 (26 to 29) | 26 (24 to 25) | 0.2443 |
| Type of surgery | | | ns |
| Wedge resection | 8 (44) | 14 (58) | |
| Segmentectomy | 5 (28) | 1 (4) | |
| Lobectomy | 5 (28) | 8 (33) | |
| Other | 0 | 1 (4) | |
| Thoracoscopy/Thoracotomy | 14/4 (78/22) | 18/6 (75/25) | 0.9991 |
| Conversion to open surgery | 0 | 2 (8) | 0.4983 |
| History of smoking* | | | 0.8277 |
| Non-smoker | 5 (31) | 6 (26) | |
| Previous smoker | 9 (56) | 12 (52) | |
| Active smoker | 2 (13) | 5 (22) | |
| Preoperative lungfunction (FEV1, | 2.6 (2.1 to 3.0) | 2.1 (1.9 to 2.4) | 0.0629 |
| L)** | | | |
| Previous lung surgery | 0 (0) | 2 (8) | 0.4983 |
| Comorbidities | | | ns |
| Asthma | 2 (11) | 0 | |
| COPD | 3 (17) | 4 (17) | |
| Hypertension | 9 (50) | 12 (50) | |
| Cong heart failure | 2 (11) | 1 (4) | |
| Cancer | 12 (67) | 11 (45) | |
| Diabetes mellitus | 2 (11) | 3 (13) | |
| Renal impairment | 1 (6) | 0 | |
| Surgical bleeding (ml), median | 0 (0-50) | 0 (0-100) | 0.762 |
| (range) | | | |
| Intraoperative ventilation settings§ | | | |
| (no,%) | | | |
| PRVC/VC/PC | 17/1/0 | 17/7/0 | 0.1257 |
| FiO2 | 69 (63 to 74) | 67.5 (73 to 72) | 0.9563 |
| PEEP (cm H <sub>2</sub> O) | 5.2 (5.2 to 5.8) | 5.5 (5.1 to 5.9) | 0.4782 |
| Ppeak (cm H <sub>2</sub> O) | 17 (16 to 19) | 18 (17 to 20) | 0.4898 |

Categorical data is presented as N (%) and continuous data as mean (95% CI) or otherwise specified. \*2 unknown in CXR arm and 1 unknown in LUS arm. \*\*1 missing value in CXR arm and 2 missing values in LUS arm. § Ventilation settings at the end of surgery on double lung ventilation, PRVC; pressure regulated volume controlled mode: VC; volume controlled mode: PC; pressure controlled mode

**Statistical analysis:** Independent t-test with Welch's correction or Mann-Whitney Utest for continuous samples. Chi-square or Fisher exact test for categorical variables.

| Outcomes | LUS (N=18) | CXR (N=24) | |
|---|---|---|---|
| No. x-rays performed per pt. | 1 (1 - 5) | 2 (1 - 6) | 0.0580 |
| Additional x-rays§ per pt. No. (%) of pts receiving additional x-rays | 0 (0 - 4)<br>4 (22%) | 0 (0 - 4)<br>8 (33%) | 0.4846<br>RR 0.80 (0.49 to<br>1.47) |
| Time to drain removal (min) | 320 (88-7709) | 315 (153-<br>9930) | 0.9150 |
| Late drain removal, >1 day (no.%) | 4 (22%) | 5 (21%) | 0.9999<br>RR 1.0 (0.60 to<br>2.3) |
| Adverse events/PPC, no. % | 7 (39%) | 6 (25%) | 0.9284<br>RR 1.35 (0.76 to<br>2.80) |
| Length of stay (days) | 4 (2-8) | 4 (3-9) | 0.2311 |

Data presented as median (range) or otherwise specified. § No of CXR performed in addition to protocol. Relative risk (95%CI) of receiving CXR in addition to protocol (1 CXR for all patients in LUS arm and 2 for lobectomies/segmentectomies and 1 for wedge resections in CXR arm). Early X-ray 4 pts in LUS arm and 6 pts in CXR arm.

**Statistical analysis:** Independent sample median test, Pearson chi square with Yates continuity correction, Mann-Whitney U test

## INTEROBSERVER AGREEMENT

Interobserver reliability for the LUS investigations, using intraclass correlation (ICC) for consistency(C) and absolute agreement (A), was evaluated for the following assessments:

Aeration score ICC-C 0.865/0.852 ICC-A 0.860/0.834 (dx/sin) Pneumothorax-ICC-C 0.883/0.809 ICC-A 0.885/0.809 (dx/sin) Pleural effusion ICC-C 0.887/0.769 ICC-A 0.882/0.776 (dx/sin) (LUS investigation no 1 in all cases)

ICC: (>0.75 good >0.8 very good >0.9 excellent)

## **SUMMARY:**

- 42 patients were included in this interim analysis, 18 in the LUS/intervention arm and 24 in the CXR arm. The trial is set to include 110 patients.
- More patients in the LUS arm were excluded due to re-scheduling of surgery, this can pose a problem as the LUS/intervention arm is more logistically demanding.

- There were no differences in baseline characteristics between patients allocated to the LUS/intervention and the CXR arm.
- There was a tendency towards lower total number of chest x-rays in the LUS/intervention group. However, this difference was smaller when looking at additional x-rays.
- There were no signals of delayed drain removal, increased number of adverse events, increased length of stay or increased number of additional x rays in the LUS/intervention arm.
- Interobserver consistency and agreement for LUS was generally very good for key assessments.